CLINICAL TRIAL: NCT02120248
Title: The Effect of Varied Intensities of Breastfeeding Peer Support on Duration of Breastfeeding Among Oregon WIC Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon WIC Program (Other Government)
Collaborators: USDA Food and Nutrition Service (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Reeder, Senior Research Analyst, Oregon WIC Program
Allocation: Randomized | Model: Single Group | Purpose: Prevention
Other Study IDs: FY04 WIC Special Project Grant
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Breastfeeding
Keywords: WIC; Oregon; Breastfeeding; Peer Counseling; Exclusive Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Participants receive standard WIC breastfeeding support but do not have contact with a breastfeeding peer counselor
- Low Intensity (Other): Participants will receive four scheduled phone calls from a peer counselor. Two prenatal calls and 2 postpartum.
  Interventions: Other: Telephone-based breastfeeding peer counseling
- High Intensity (Active Comparator): Participants will receive eight scheduled phone contacts from a peer counselor. Two are prenatal and 6 are postpartum.
  Interventions: Other: Telephone-based breastfeeding peer counseling

INTERVENTIONS:
Other: Telephone-based breastfeeding peer counseling
  Arms: High Intensity; Low Intensity

SUMMARY:
The U.S. Surgeon General has recommended that peer counseling to support breastfeeding become a core service of the Supplemental Nutrition Program for Women, Infants and Children (WIC). As of 2008, 50 percent of WIC clients received services from local WIC agencies that offered peer counseling. Little is known as to the effectiveness of these peer counseling programs. Randomized controlled trials of peer counseling interventions among low-income women in the U.S. showed increases in breastfeeding initiation and duration, but it is doubtful that the level of support provided could be scaled up to service WIC clients nationally. The investigators tested whether a telephone peer counseling program among WIC participants could increase breastfeeding initiation, duration and exclusivity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Oregon WIC participants in Jackson, Washington and Hood River counties or Umatilla Morrow Head Start.

Exclusion Criteria:

* WIC participant outside of the 4 study agencies.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1948 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 6 months postpartum

SECONDARY OUTCOMES:
Exclusive breastfeeding | 3 months postpartum

OTHER OUTCOMES:
Partial Breastfeeding | 3 months
Partial breastfeeding | 6 months postpartum

REFERENCES:
- [Derived] Reeder JA, Joyce T, Sibley K, Arnold D, Altindag O. Telephone peer counseling of breastfeeding among WIC participants: a randomized controlled trial. Pediatrics. 2014 Sep;134(3):e700-9. doi: 10.1542/peds.2013-4146. Epub 2014 Aug 4. PMID 25092936